CLINICAL TRIAL: NCT02275559
Title: Asthma Symptom Management Through Mindfulness Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: The Miriam Hospital (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Lori Pbert, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H00006718; R01AT008393 (NIH)
Record Dates: First submitted 2014-10-06; First posted 2014-10-27 (Estimated); Results first posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): Mindfulness Based Stress Reduction (MBSR) program consists of 8 weekly classes plus an all-day class to train participants in mindfulness and its application, including addressing challenges arising from chronic diseases and life stresses.
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR)
- Healthy Living Course (HLC) (Active Comparator): The Healthy Living Course (HLC) consists of 8 weekly classes plus an all-day class providing lectures and discussions about health-related topics. The purpose of the HLC is to match the MBSR for time, attention and group support
  Interventions: Behavioral: Healthy Living Course (HLC)

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) — Mindfulness Based Stress Reduction (MBSR) program consists of 8 weekly classes plus an all-day class to train participants in mindfulness and its application, including addressing challenges arising from chronic diseases and life stresses.
  Arms: Mindfulness Based Stress Reduction
Behavioral: Healthy Living Course (HLC) — The Healthy Living Course (HLC) consists of 8 weekly classes plus an all-day class providing lectures and discussions about health-related topics. The purpose of the HLC is to match the MBSR for time, attention and group support
  Arms: Healthy Living Course (HLC)

SUMMARY:
Asthma is one of the four most common adult chronic disorders. Supporting asthma patients in improving their asthma control and symptoms as well as their quality of life are important goals in clinical management. This study will test the effect of a widely-available mindfulness training program in improving asthma control and symptoms and quality of life among patients with asthma, and explore the relationship between asthma control and a number of factors, including how well patients perceive their respiratory symptoms.

DETAILED DESCRIPTION:
Asthma is one of the four most common adult chronic disorders. It affects 7.3% (16.4 million) U.S. adults and costs $18 billion in direct healthcare costs and lost productivity. Control of symptoms and improving patient's quality of life (QOL) are the goals in asthma management and require patients to accurately identify their symptoms. But the low congruence between patients' symptom reports and their pulmonary function leads to disease management errors. The accuracy with which asthma patients recognize their symptoms is affected by emotional factors, and because high negative affectivity is related to low interoceptive accuracy and worse asthma symptoms and asthma physical health, the frequent mental distress prevalent among asthmatics is thought to result in difficulty in distinguishing symptoms of stress/distress from those of asthma. Mindfulness training teaches people to recognize and distinguish among the components of experience (thoughts, feelings, sensations/symptoms) and is associated with increased perceptual accuracy of respiratory resistance, and reduced affective negativity. It thus has the potential to improve patient's discrimination between asthma symptoms and stress/distress, resulting in improved asthma management, control and QOL. A pilot randomized controlled trial (RCT) (N=84) of a widely-available mindfulness training program (Mindfulness-Based Stress Reduction (MBSR)) to explore this hypothesis in adults with mild, moderate or severe persistent asthma. Intent to treat analyses comparing MBSR to an active control program showed clinically significant improvements in overall QOL (p=0.01), as well as important improvements in asthma symptoms (p=0.009), reduced use of asthma rescue medication (p=0.001), anxiety (p=0.05), perceived stress (p=0.01), and mindfulness (p=0.01). Promising improvements in the percentage of patients with well-controlled asthma also were found. All improvements were sustained 10 months post-intervention. Widespread adoption of this promising adjunct intervention will require sharper evidence regarding asthma control and symptoms. The primary aim is to test MBSR against an active control on the key clinical outcomes of asthma control and symptoms using gold standard measures with 256 adults with mild, moderate or severe asthma. And to evaluate the program's effect on asthma QOL, lung function, cost-effectiveness, and the mediating effect of respiratory interoceptive accuracy on asthma control, QOL, and medication use. Assessments are at baseline, 6-, 12-, and 18-month follow-up. MBSR is available nationwide and covered by many third-party payers. If sustained and credible improvements in asthma control and symptoms are found, MBSR could be a useful adjunct to traditional medical treatment and would have the potential for improving the lives of people with asthma. By examining the mediating effects of psychosocial variables on asthma control, the study also generates new knowledge on mechanisms of change and maintenance in mind-body and behavioral programs in medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Documented diagnosis of asthma from a physician for greater than 12 months that includes an objective indicator of bronchial hyperresponsiveness (positive methacholine challenge test or > 12% improvement in forced expiratory volume in 1 second (FEV1) or forced vital capacity (FVC) in response to bronchodilator);
* Meets criteria for mild, moderate or severe asthma
* Treatment with inhaled corticosteroids for at least 12 weeks with stable dosing for greater than 4 weeks;
* Able to read and understand English, and complete informed consent process and study data collection procedures.

Exclusion Criteria:

* Current smoker or greater than 10 pack-year smoking history
* Diagnosis of asthma of intermittent severity
* Other lung diseases besides asthma
* Cancer, except non-melanoma skin cancer;
* Currently receiving treatment for symptomatic cardiovascular disease within past 6 months
* Current or recent (within the past 3 months) severe exacerbation of asthma requiring hospitalization or oral glucocorticoids;
* Currently pregnant
* Major psychiatric disorders or psychiatric hospitalization in the last 2 years;
* Has taken the MBSR program in the past, and/or currently practicing meditation or yoga on a regular basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Carmody, PhD, Principal Investigator — University of Massachusetts, Worcester; Lori Pbert, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction | Healthy Living Course (HLC)
Started | 115 | 118
Completed | 115 | 118
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction | Healthy Living Course (HLC) | Total
Number analyzed (Participants) | 115 | 118 | 233
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.72 (12.69) | 51.96 (14.75) | 52.84 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 97 | 194
  Male | 18 | 21 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 16 | 26
  White | 91 | 92 | 183
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 10 | 24
Region of Enrollment [Number; unit: participants] — Two sites; Rhode Island and Massachusetts.
  participants
    United States | 115 | 118 | 233

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Asthma Control at 18 Months
Description: Asthma control will be assessed using the Asthma Control Questionnaire (ACQ). The ACQ is a 7-item validated measure that assesses the 5 asthma symptoms considered most important and most used by clinicians for evaluating asthma control, along with use of short-acting beta-agonist and FEV1 percent predicted. Patients recall their symptoms and short-acting beta-agonist use during the previous week; FEV1 is obtained from spirometry. All seven questions are scored on a 7-point scale (0=good control, 6=poor control), and the overall score (range 0-6) is the mean of the seven responses. Lower scores indicate better outcome. Minimum = 0, Maximum = 6. Changes of 0.5 or greater in the score are considered important differences.
Time Frame: Baseline and 18 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Healthy Living Course (HLC)
Number analyzed (Participants) | 101 | 106
score on a scale | 1.27 (0.11) | 1.17 (0.09)

2. Secondary Outcome: Change From Baseline in Asthma-related Quality of Life at 18 Months
Description: Asthma-related quality of life will be assessed using the Asthma-related QoL (AQoL) measure.The AQoL has 30 items assessing impairment in 4 areas of function shown to be important to the QoL of adult patients with asthma (activity limitations, asthma symptoms, emotional function and environmental exposure). Overall QoL is computed by averaging scores on the 4 domains. Items assess the degree to which important activities have been limited by asthma during the last 2 weeks on a 7-point scale (1= maximal impairment, 7= no impairment). Shown to be valid, reliable and sufficiently sensitive to changes in asthma symptoms to capture the effects of an intervention in a clinical trial. Higher scores = better outcome, minimum score = 30, maximum score 210. Changes in scores of 0.5 or above represent clinically meaningful improvement in QoL.
Time Frame: Baseline and 18 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Healthy Living Course (HLC)
Number analyzed (Participants) | 99 | 106
score on a scale | 5.19 (0.13) | 5.29 (0.11)

3. Secondary Outcome: Change From Baseline in Respiratory Interoceptive Accuracy at 18-months
Description: Respiratory interoceptive accuracy will be measured using the Breath Perception Discrimination Test (BPDT). The BPDT measures ability to detect small changes in resistive load. This test will be done in the Pulmonary Diagnostic Laboratory at each site. During the test period, the presentation of the resistor will be announced at the onset of a new inspiration for the duration of one full breath cycle. At the conclusion of the breath cycle, participants pause for 5 normal breaths, at which point the next resistor in the block is presented. The test will be divided into 6 blocks during which there is a random presentation of each resistor so that participants carry out 30 ratings (6 for each condition) over the course of the test. Higher score is better outcome, lower score is worse outcome. Lowest score is zero percent, highest score is 100% Time to complete: 30 minutes.
Time Frame: Baseline and 18-months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Healthy Living Course (HLC)
Number analyzed (Participants) | 68 | 73
score on a scale | 0.79 (0.01) | 0.77 (0.01)

4. Secondary Outcome: Change From Baseline in Percent Predicted Expiratory Volume at 18-months.
Description: Lung function will be assessed via spirometry. Spirometry assesses the level of air flow limitation according to the forced expiratory volume in 1 second (FEV1). The unit of measure is not a score on a scale but rather "percent predicted expiratory volume" to assess air flow limitation. Measurement will be done in the site Pulmonary Diagnostic Laboratories according to American Thoracic Society guidelines before and after inhalation of bronchodilator. This includes instructing participants to not take a bronchodilator at least 4 hours prior to their spirometry, and assessing lung function both before, and then 30 minutes after bronchodilator to assess best lung function and responsiveness to bronchodilator therapy. Higher scores mean better outcome.
Time Frame: Baseline and 18-months
Population: This combination of the two arms was the prespecified analysis.
Measure: Mean (Standard Error); unit: percent predicted expiratory volume
Arm/Group | Mindfulness Based Stress Reduction | Healthy Living Course (HLC)
Number analyzed (Participants) | 71 | 65
percent predicted expiratory volume | 360.89 (8.92) | 351.8 (12.07)

5. Secondary Outcome: Cost Per Change in Quality of Life (QOL)
Description: This outcome is the Incremental Cost Effectiveness Ratio (ICER). The ICER estimates how much the MBSR intervention costs, relative to the HLC intervention, to improve the outcome measure by 1 unit. The ICER is calculated by dividing the incremental cost by the incremental outcome. The Incremental cost is difference in total costs (sum of program costs and healthcare costs over 18 months, in U.S. dollars) between the MBSR and HLC groups. The Incremental outcome is the difference between the groups in the chosen measure of health outcome at 18 months (here, mean Asthma-related QoL (AQoL) questionnaire scores).
Time Frame: 18 months
Population: This combination of the two arms was the prespecified analysis.
Measure: Number; unit: U.S. Dollars/1 point of QOL improvement
Groups:
- Mindfulness Based Stress Reduction Compared to Healthy Living Course: Mindfulness Based Stress Reduction (MBSR) program consists of 8 weekly classes plus an all-day class to train participants in mindfulness and its application, including addressing challenges arising from chronic diseases and life stresses.
  The Healthy Living Course (HLC) consists of 8 weekly classes plus an all-day class providing lectures and discussions about health-related topics. The purpose of the HLC is to match the MBSR for time, attention and group support
  The two arms are combined for this analysis
Arm/Group | Mindfulness Based Stress Reduction Compared to Healthy Living Course
Number analyzed (Participants) | 233
U.S. Dollars/1 point of QOL improvement | 10,006

6. Secondary Outcome: Cost in Change of Percent Predicted FEV
Description: This outcome is the Incremental Cost Effectiveness Ratio (ICER). The ICER estimates how much the MBSR intervention costs, relative to the HL intervention, to improve the outcome measure by 1 unit. The ICER is calculated by dividing the incremental cost by the incremental outcome. The incremental cost is the difference in total costs (sum of program costs and healthcare costs over 18 months, in U.S. dollars) between the MBSR and HLC groups. The incremental outcome is the difference between the groups at 18 months in the chosen measure of health outcome (here, mean Predicted FEV1 scores). This is not a scale.
Time Frame: 18 months
Population: This combination of the two arms was the prespecified analysis.
Measure: Number; unit: US. Dollars/1 point % Predicted FEV
Groups:
- Mindfulness Based Stress Reduction Compared to Healthy Living Course: Mindfulness Based Stress Reduction (MBSR) program consists of 8 weekly classes plus an all-day class to train participants in mindfulness and its application, including addressing challenges arising from chronic diseases and life stresses.
  Healthy Living Course (HLC): The Healthy Living Course (HLC) consists of 8 weekly classes plus an all-day class providing lectures and discussions about health-related topics. The purpose of the HLC is to match the MBSR for time, attention and group support
  The two arms are combined for this analysis
Arm/Group | Mindfulness Based Stress Reduction Compared to Healthy Living Course
Number analyzed (Participants) | 233
US. Dollars/1 point % Predicted FEV | 145

7. Secondary Outcome: Cost in Change of Asthma Control
Description: This outcome is the Incremental Cost Effectiveness Ratio (ICER). The ICER estimates how much the MBSR intervention costs, relative to the HL intervention, to improve the outcome measure by 1 unit. The ICER is calculated by dividing the Incremental cost by the incremental outcome. The incremental cost is the difference in total costs (sum of program costs and healthcare costs over 18 months, in U.S. dollars) between the MBSR and HLC groups. The incremental outcome is the difference between the groups in the chosen measure of health outcome 18 months (here, mean Asthma Control Score). This is not a scale.
Time Frame: 18 months
Population: This combination of the two arms was the prespecified analysis.
Measure: Number; unit: US $/1 point of Change of Asthma Control
Arm/Group | Mindfulness Based Stress Reduction Compared to Healthy Living Course
Number analyzed (Participants) | 233
US $/1 point of Change of Asthma Control | 3,255

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Mindfulness Based Stress Reduction | Healthy Living Course (HLC)
All-Cause Mortality (participants affected / at risk) | 0/115 | 1/118
Serious Adverse Events (participants affected / at risk) | 12/115 | 18/118
Other Adverse Events (participants affected / at risk) | 10/115 | 10/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Stress Reduction (N=115) | Healthy Living Course (HLC) (N=118)
Bilateral lower extremity pain with weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Inpatient hospitalization with subsequent adult partial program admission (Psychiatric disorders) | 1 (1) | 0 (0)
Chest congestion associated with l sided arm weakness and lower extremity weakness & numbness (Cardiac disorders) | 1 (1) | 0 (0)
Surgical repair of lumbar spondylosis with radiculopathy (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 4 (4) | 0 (0)
Kidney Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Appendectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Microcytic anemia with iron deficiency, secondary to gi blood loss in the setting of nsaid use (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Thyroid Gland Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Dysphagia & dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Emphysematous pyelonephritis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia due to infectious organism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Broken hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Surgery; L4/5 discectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Peritoneal abscess (Gastrointestinal disorders) | 0 (0) | 1 (1)
Recurrent major depressive episode (Psychiatric disorders) | 0 (0) | 1 (1)
Drug-induced, allergic reaction to Bactrim (Infections and infestations) | 0 (0) | 1 (1)
Arthritis spinal stenosis and spondylolisthesis surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgery to repair small bowel obstruction (Surgical and medical procedures) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Hernia Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Abdominal myomectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Chest pain & syncope (Cardiac disorders) | 0 (0) | 1 (1)
Slurred speech ruled out TIA (Nervous system disorders) | 0 (0) | 1 (1)
Patient fell (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Stress Reduction (N=115) | Healthy Living Course (HLC) (N=118)
Clinically significant decrease of ≥ 15% in spirometry from baseline in FEV1. (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT02275559/Prot_SAP_001.pdf
  • Informed Consent Form (2018-06-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT02275559/ICF_000.pdf